CLINICAL TRIAL: NCT06562738
Title: Clinical Study on Efficacy and Safety of Hetrombopag in the Preoperative Patients of Thrombocytopenia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Third People's Hospital of Chengdu (Other)
Collaborators: Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Principal Investigator, Ying Li, Principal Investigator, The Third People's Hospital of Chengdu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ThirdHospitalChengdu
Record Dates: First submitted 2024-08-13; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Thrombocytopenia
Keywords: Hetrombopag; Thrombocytopenia; Preoperative
MeSH Terms: conditions — Thrombocytopenia | interventions — hetrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Hetrombopag arm (Experimental): Takes Hetrombopag 7.5 mg/day at bedtime for at most 14 days.
  Interventions: Drug: Hetrombopag

INTERVENTIONS:
Drug: Hetrombopag — Hetrombopag 7.5 mg, once a day, at bedtime for up to 14 days, drug administration was stopped when PLT≥100 ×10^9/L, and take blood routine examination weekly, drug administration was resumed when PLT < 100 ×10^9/L. When PLT ≤30× 10^9/L or ≥300 ×10^9/L, take blood routine examination every 3 days.

SUMMARY:
This is an investigator-initiated, single-arm, prospective clinical study to evaluate the efficacy and safety of heptapopal in the treatment of thrombocytopenia prior to elective surgery

DETAILED DESCRIPTION:
It was planned to include 55 patients with immune thrombocytopenia with preoperative platelet ≤75×10^9/L. After signing the informed consent letter, the patients will enter the screening period (up to 7 days), and after passing the screening, they will receive oral hexapopal treatment, the specific medication regimen is: 7.5mg, once a day, taken orally on an empty stomach before going to bed, for a maximum of 14 days, and stop the drug when PLT≥100×10^9/L. During the oral administration of hexapopal, the administration was suspended when PLT≥200×10^9/L, and continued when the blood image was monitored weekly until PLT < 100×10^9/L. During the treatment period, blood routine was monitored every 7 days, and when PLT≤30×10^9/L or ≥300×10^9/L, blood routine was monitored every 3 days. Patients will have an end-of-treatment visit within 7 days of stopping treatment, followed by a 30-day safe follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old; diagnosis of immune thrombocytopenia.
2. Platelets ≤75×10^9/L before scheduled elective surgery.

Exclusion Criteria:

1. History of allergy to Thrombopoietin Receptor Agonists (TPO-RA) drugs;
2. Severe bleeding symptoms, such as gastrointestinal bleeding, bleeding of important organs, and intracranial bleeding;
3. Thrombotic diseases, such as pulmonary embolism, arterial thrombosis and disseminated intravascular coagulation (DIC);
4. Positive anti-human immunodeficiency virus antibody or anti-treponema pallidum specific antibody;
5. New York Heart Association (NYHA) Grade 3 or 4 congestive heart failure;
6. History of angina pectoris, myocardial infarction or cerebral infarction within 6 months before the screening period;
7. Have an active infection that is difficult to control;
8. Pregnant or lactating women;
9. Other conditions determined by the investigator to be unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Platelet elevation | up to 14 days
  Proportion of patients achieving perioperative platelet count goals (≥80×10^9/ L for major surgery and ≥50×10^9/ L for minor surgery) without emergency treatment

SECONDARY OUTCOMES:
Secondary Outcome | up to 14 days
  The median time to reach the platelet count target;

CONTACTS AND LOCATIONS:
Overall Officials: JING TAN, MD, Principal Investigator — 成都市第三人民医院
Locations (1):
- Chengdu Third People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

DOCUMENTS (2):
  • Study Protocol (2023-12-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT06562738/Prot_000.pdf
  • Informed Consent Form (2023-12-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT06562738/ICF_001.pdf